CLINICAL TRIAL: NCT02030587
Title: Laparoscopic Adrenalectomy Versus Radiofrequency Ablation for Aldosterone-producing Adenoma: a Prospective Randomized Controlled Trial
Brief Title: Laparoscopic Adrenalectomy Versus Radiofrequency Ablation
Acronym: LARFA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Enders K.W. Ng, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2012.193-T
Record Dates: First submitted 2014-01-05; First posted 2014-01-08 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Hyperaldosteronism; Conn Syndrome; Adrenocortical Adenoma
Keywords: Hyperaldosteronism; Adrenocortical adenoma; Adrenalectomy; Catheter ablation
MeSH Terms: conditions — Hyperaldosteronism; Adrenocortical Adenoma | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiofrequency Ablation (Experimental): Radiofrequency Ablation
  Interventions: Procedure: Radiofrequency Ablation
- Laparoscopic Adrenalectomy (Active Comparator): Laparoscopic Adrenalectomy
  Interventions: Procedure: Laparoscopic Adrenalectomy

INTERVENTIONS:
Procedure: Radiofrequency Ablation
  Arms: Radiofrequency Ablation
Procedure: Laparoscopic Adrenalectomy
  Arms: Laparoscopic Adrenalectomy

SUMMARY:
This is a prospective randomized controlled study comparing laparoscopic adrenalectomy (LA) versus image-guided percutaneous radiofrequency ablation (RFA) in treating aldosterone-producing adenoma.

The objectives of this study are to

1. compare the short-term outcomes of LA and RFA in treating aldosterone-producing adenoma.
2. compare the treatment success rates of LA and RFA during follow-up for primary aldosteronism.

ELIGIBILITY:
Inclusion Criteria:

1. Hypertensive individuals
2. Biochemically confirmed primary aldosteronism
3. Radiologically confirmed unilateral adrenal adenoma ≤3cm

Exclusion Criteria:

1. Bilateral adrenal disease
2. Multiple adrenal tumors
3. Other concomitant adrenal diseases
4. Potentially malignant adrenal tumors as shown on imaging
5. Uncorrected coagulopathy
6. Surgically unfit for general anaesthesia
7. Prior open abdominal surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-01; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Morbidity rate | 30-day
Resolution of hyperaldosteronism | 1 year

SECONDARY OUTCOMES:
Operative time | 24 hours
Periprocedural hypertensive crisis | 24 hours
Mortality rate | 30 days
Blood loss | 24 hours
Analgesic requirement | 30 days
Time to resumption of activity | 30 days
Resolution of hypokalaemia | 1 year
Blood pressure control | 1 year
Hospital stay | 30 days
Pain score | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Enders KW Ng, MB ChB, Study Chair — Chinese University of Hong Kong; Shirley YW Liu, MB ChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

REFERENCES:
- [Background] Liu SY, Ng EK, Lee PS, Wong SK, Chiu PW, Mui WL, So WY, Chow FC. Radiofrequency ablation for benign aldosterone-producing adenoma: a scarless technique to an old disease. Ann Surg. 2010 Dec;252(6):1058-64. doi: 10.1097/SLA.0b013e318f66936. PMID 21107117